CLINICAL TRIAL: NCT04078178
Title: A Crossover, Randomized Block Sequence, Double-Blind, Placebo-Controlled Trial for Nicotinamide Riboside in Subjective Cognitive Decline and Mild Cognitive Impairment in Aging
Brief Title: Crossover Trial for Nicotinamide Riboside in Subjective Cognitive Decline and Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven E Arnold, MD (Other)
Responsible Party: Sponsor-Investigator, Steven E Arnold, MD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2019P002668
Record Dates: First submitted 2019-08-27; First posted 2019-09-04 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Cognition Disorders in Old Age; Mild Cognitive Impairment; Cognitive Decline
Keywords: Mild Cognitiive Impairment; Subjective Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Participants were randomized into 2 Treatment sequences, one starting with Placebo followed by Niagen; and the other sequence starting with Active Niagen and followed by Placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Active Niagen, Placebo (Experimental): Subjects received 1000 mg Niagen and PBO dispensed in randomized blocks. Participants in Sequence 1 took Niagen daily for 8 weeks, followed by Placebo daily for 8 weeks.
  Interventions: Dietary Supplement: Niagen; Dietary Supplement: Placebo Comparator
- Sequence 2: Placebo, Active Niagen (Experimental): Subjects received 1000 mg Niagen and PBO dispensed in randomized blocks. Participants in Sequence 2 took Placebo daily for 8 weeks, followed by Active Niagen daily for 8 weeks.
  Interventions: Dietary Supplement: Niagen; Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Niagen — Nicotinamide Riboside
Dietary Supplement: Placebo Comparator — Placebo

SUMMARY:
In this research study we want to learn more about whether taking Niagen, a daily supplement containing a form of Vitamin B3, will improve cognitive function, mood, and daily activity in people with Subjective Cognitive Decline (SCD) or Mild Cognitive Impairment (MCI).

DETAILED DESCRIPTION:
Over a 6 month period, we will ask study participants to take both Niagen or a placebo for 8 weeks each and complete research visits ever 4 or 8 weeks. Most research visits will involve a blood draw, cognitive testing, and mood questionnaires. We will ask you to come to our center 4-5 times to complete some study activities in-person. There will be an option to participate in a lumbar puncture sub-study, in which participants would have up to 3 lumbar punctures. There will also be an option to participate in an MRI sub-study, in which participants would have up to 3 MRIs over the course of the study. In between research visits, we will also ask the participants to wear a Fitbit activity tracker and play computerized brain games a few times a week. This will enable us to get a snapshot of each subject's functioning levels day to day and better determine whether or not the supplement is having an effect on the participant.

ELIGIBILITY:
Inclusion criteria:

1. Ages 60 and up;
2. Memory and other cognitive complaints consistent with SCD or MCI as defined by the National Institute on Aging:

   a. SCD will be defined as: i. any subjective concern of change in cognitive functioning without objective evidence of cognitive impairment, and ii. complete preservation of functional abilities and independence in instrumental activities of daily living.

   b. MCI will be defined as: i. a preexisting diagnosis of MCI given by a trained physician or behavioral health provider, or ii. evidence of objective impairment in cognitive functioning in one or more domain with preservation of functional abilities and independence in instrumental activities of daily living as defined by the National Institute on Aging;
3. Minimum score of 16 on t-MoCA;
4. Ability to provide direct informed consent as assessed by obtaining a score of 70% on questions 1-10, and answer 'yes' to questions 11-14 of the Informed Consent Worksheet after two attempts;
5. Education level, English language skills and literacy indicates participant able to complete all assessments;
6. Willing and able to complete all assessment and study procedures;
7. Not pregnant, lactating, or of child-bearing potential;
8. If on cholinesterase inhibitor and/or memantine, doses are stable for 3 months prior to baseline.

Exclusion Criteria:

1. Any specific CNS disease history other than suspected ADRD, such as major clinical stroke, brain tumor, normal pressure hydrocephalus, multiple sclerosis, significant head trauma with persistent neurological of cognitive deficits or complaints;
2. Any impairment in instrumental activities of daily living that would indicate a level of cognitive impairment beyond MCI as assessed by a trained rater;
3. Clinically significant unstable medical condition that could affect safety or compliance with the study and would, in the opinion of the investigator, pose a risk to the participant if they were to participate in the study;
4. History of neuroimaging with evidence of major infarction, injury, infection, or other focal lesions that may be related to cognitive dysfunction;
5. If participating in the optional lumbar puncture sub-study, any contraindication to undergo lumbar punctures, such as:

   1. abnormal coagulation PT/INR test result, outside of the normal range of 0.9 to 1.2 platelet counts below 50,000 (determined by a licensed study physician or Nurse Practitioner after reading test results).
   2. Platelet counts below 50,000.
   3. Use of Coumadin, Warfarin, or other blood thinner medications.
   4. Infection near the puncture site, or spinal column deformities (a licensed physician or Nurse Practitioner will examine the site visually for infection or spinal deformities before performing the procedure).
   5. Known allergy to Lidocaine.
6. Major active or chronic unstable psychiatric illness (e.g. depression, bipolar disorder, obsessive compulsive disorder, schizophrenia) within the previous year;
7. Current suicidal ideation or history of suicide attempt;
8. History of alcohol or other substance abuse or dependence within the past two years;
9. Any significant systemic illness or medical condition that could affect safety or compliance with study;
10. Laboratory abnormalities in Vitamin B12, Thyroid Stimulating Hormone (TSH), or other common laboratory parameters that might contribute to cognitive dysfunction or other abnormalities in hematological, hepatic or renal function tests;
11. Current use of medications with psychoactive properties that in the opinion of the principal investigator, may be deleteriously affecting cognition (e.g., anticholinergics, antihistamines, antipsychotics, sedative hypnotics, anxiolytics);
12. Any known hypersensitivity to nicotinamide riboside, or its principal metabolite, nicotinamide mononucleotide;
13. No consumption of dietary supplements containing more than 100mg niacin, nicotinamide riboside (NR), or nicotinamide mononucleotide (NMN) as the primary agents 30 days prior to baseline and for the duration of the trial;
14. Use of other investigational agents or interventions one month prior to entry and for the duration of the trial;
15. If participating in the optional MR sub-study: Any contraindication to undergo MRI studies, such as history of cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head, prosthetic heart valves, and/or severe claustrophobia impeding ability to participate in an imaging study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Arnold, MD, Principal Investigator — MGH
Locations (1):
- Alzheimer's Clinical and Translational Research Unit, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
All data will be DE-Identified

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 61 Participants signed consent and enrolled in the study. Prior to randomization assignment, 15 participants screen failed. 46 proceeded to randomization assignment and study lead-in.
Groups:
- Sequence 1: Niagen, Then Placebo: Subjects received 1000 mg Niagen daily for 8 weeks. After 8 weeks of Niagen, participants took Placebo daily for 8 weeks.
  Niagen: Nicotinamide Riboside
- Sequence 2: Placebo, Then Niagen: Subjects received Placebo daily for 8 weeks, then participants received 1000mg Active Niagen daily for 8 weeks.
  Niagen: Nicotinamide Riboside
Period: Lead-In Period (4-Weeks)
Arm/Group | Sequence 1: Niagen, Then Placebo | Sequence 2: Placebo, Then Niagen
Started | 23 | 23
Completed | 22 | 20
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Screen Fail | 1 | 2
Period: Baseline/Initial Treatment (8 Weeks)
Arm/Group | Sequence 1: Niagen, Then Placebo | Sequence 2: Placebo, Then Niagen
Started | 22 | 20
Completed | 20 | 18
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Early Termination | 1 | 0
Period: Crossover Treatment (8 Weeks)
Arm/Group | Sequence 1: Niagen, Then Placebo | Sequence 2: Placebo, Then Niagen
Started | 20 | 18
Completed | 20 | 17
Not Completed | 0 | 1
Not completed — Early Termination | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Active Niagen, Placebo | Sequence 2: Placebo, Active Niagen | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 16 | 11 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 17 | 37
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Niagen vs PBO on Cognition as Measured by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
Description: The primary outcome of this study will be objective measures of cognitive performance measured with the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) at baseline, crossover, and the end of study. RBANS has a mean score of 100 with a standard deviation of 15. Scores range from 40 to 160. Higher scores indicate normal cognition.
Time Frame: From baseline through end of study at 16 weeks
Population: Participants that completed the trial were analyzed (20 in sequence 1; 17 in sequence 2)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sequence 1: Active Niagen, Placebo | Sequence 2: Placebo, Active Niagen
Number analyzed (Participants) | 20 | 17
units on a scale
  Baseline | 92.15 (2.68) | 91.04 (3.15)
  1st intervention/crossover 8 weeks | 94.87 (2.68) | 95.17 (3.16)
  16 weeks/end of study | 93 (3.1) | 95.64 (3.58)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant from the baseline visit to end of study, 20 weeks. In the NR-Placebo group (Sequence 1), there were 22 participants that started Baseline, with 2 withdrawing/Early Termination before crossover. In the Placebo- NR group (Sequence 2), there were 20 participants that started baseline (Placebo) and then 18 who crossed over into the NR group. Data was collected for 22 participants in Sequence 1 and 20 participants in Sequence 2.
Groups:
- Sequence 1: Baseline (Niagen); Sequence 1: Crossover (Placebo): Subjects received 1000 mg Niagen and PBO dispensed in randomized blocks. Participants in Sequence 1 took Niagen daily for 8 weeks, followed by Placebo daily for 8 weeks.
  Niagen: Nicotinamide Riboside
  Placebo Comparator: Placebo
- Sequence 2: Baseline (Placebo); Sequence 2: Crossover (Niagen): Subjects received 1000 mg Niagen and PBO dispensed in randomized blocks. Participants in Sequence 2 took Placebo daily for 8 weeks, followed by Active Niagen daily for 8 weeks.
  Niagen: Nicotinamide Riboside
  Placebo Comparator: Placebo
Arm/Group | Sequence 1: Baseline (Niagen) | Sequence 1: Crossover (Placebo) | Sequence 2: Baseline (Placebo) | Sequence 2: Crossover (Niagen)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 1/20 | 2/18
Other Adverse Events (participants affected / at risk) | 3/22 | 2/20 | 3/20 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1: Baseline (Niagen) (N=22) | Sequence 1: Crossover (Placebo) (N=20) | Sequence 2: Baseline (Placebo) (N=20) | Sequence 2: Crossover (Niagen) (N=18)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1: Baseline (Niagen) (N=22) | Sequence 1: Crossover (Placebo) (N=20) | Sequence 2: Baseline (Placebo) (N=20) | Sequence 2: Crossover (Niagen) (N=18)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cramping (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 3 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT04078178/Prot_SAP_000.pdf